CLINICAL TRIAL: NCT03153917
Title: Wake-sleep Cycle and Melatonin Secretion Dynamics Associated With 12 Hours Shift Work in French Nurses
Brief Title: Biological Rhythms Impact of 12 Hours Shift Work
Acronym: MELACTI-12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0624
Record Dates: First submitted 2017-04-20; First posted 2017-05-15 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-04

CONDITIONS: Shift-Work Sleep Disorder
Keywords: shift work; melatonin; sleep
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- melatonin and cortisol sampling (Experimental): 14 healthy volunteer nurses working on 12 hours night/day schedules in the Sleep Medicine Center of Lyon.
  Interventions: Other: melatonin and cortisol sampling

INTERVENTIONS:
Other: melatonin and cortisol sampling — The study will take place over 15 days during which the nurses will wear an actigraphic wristband and will fulfill a sleep log. During 3 periods of 24 hours selected during these 15 days, including a 12h day shift (Day 2), a 12h night shift (Day 8) and a rest (Day 13), the participants will collect their urine by 4 to 8 hour periods, note the corresponding urine volumes and for each period, sample a 5 mL tube which will be analyzed later (6-sulfatoxymelatonin and urinary cortisol assays). The subjects will complete questionnaires at the beginning of the study (Horne and Ostberg, Insomnia Severity Index, Epworth, Pichot, Hospital Anxiety and Depression) and the days corresponding to the urine sampling (Karolinska and St Mary Hospital).

SUMMARY:
Nonstandard time-schedules work are widespread in the world of work. Shift and night work have been shown to be responsible for a desynchronization of biological rhythms, associated with melatonin secretion impairment and sleep disturbances. However, while health consequences of night and shift work are widely recognized and represent a major public health concern (High Authority of Health 2012 Recommendations and National Agency for Public Health Food, Environment and Work 2016 Report), the mechanisms by which the circadian system is affected by shift work remain poorly understood. Indeed most of the studies in the fields are cross-sectional, based on few blood or urinary samples in a single work position, in workers whose shift work patterns are often misidentified and heterogeneous. Moreover, few studies have assessed melatonin secretion alterations in relation to objective sleep measurement (actigraphy). The aim of this study is to assess the dynamics of melatonin secretion adaptation in 12-hour shift work and to correlate these data to sleep-wake cycle recording.

ELIGIBILITY:
Inclusion Criteria:

* Nurses or nursing assistants working in the Sleep and Respiratory Diseases Department of the Croix-Rousse Hospital with positions in 12 hours for more than 6 months
* informed consent given by the subject

Exclusion Criteria:

* Pregnancy or lactation <6 months
* Taking treatment modifying the secretion of melatonin (melatoninergic drugs (including antidepressants), beta-blockers)
* Refusal of participate
* Minor or major protected subject
* Not affiliated to a social security scheme
* Participant in another interventional study interfering with sleep / wake rhythm or work schedules (judgment of the investigator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
total amount of melatonin excreted during the sleep period for the night shift | at day 8 (night shift)
  The impact of 12H shift work on melatonin secretion dynamics will be assessed by comparing the total amount of melatonin excreted during the sleep period between the 12h day shift condition and the 12h night shift condition
total amount of melatonin excreted during the sleep period for the day shift. | at day 2 (day shift)
  The impact of 12H shift work on melatonin secretion dynamics will be assessed by comparing the total amount of melatonin excreted during the sleep period between the 12h day shift condition and the 12h night shift condition

SECONDARY OUTCOMES:
Total amount of melatonin excreted during the sleep period at rest | at day 13 (rest)
  the total amount of melatonin excreted during the sleep period at rest will be compared to the total amount of melatonin excreted during the sleep period for the 12h day shift condition ant to the total amount of melatonin excreted during the sleep period for the 12h night shift condition
Melatonin secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Melatonin secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Melatonin secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Melatonin secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Melatonin secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Melatonin secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Melatonin secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Melatonin secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Melatonin secretion dynamics at rest | at day 13 (rest)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Melatonin secretion dynamics at rest | at day 13 (rest)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Melatonin secretion dynamics at rest | at day 13 (rest)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Melatonin secretion dynamics at rest | at day 13 (rest)
  Secretion of melatonin on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Cortisol secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Cortisol secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Cortisol secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Cortisol secretion dynamics in 12h day shift | at day 2 (day shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Cortisol secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Cortisol secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Cortisol secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Cortisol secretion dynamics in 12h night shift | at day 8 (night shift)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Cortisol secretion dynamics at rest | at day 13 (rest)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of total excretion (ng)
Cortisol secretion dynamics at rest | at day 13 (rest)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of acrophase (h)
Cortisol secretion dynamics at rest | at day 13 (rest)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of amplitude (ng)
Cortisol secretion dynamics at rest | at day 13 (rest)
  Secretion of cortisol on sequential urinary specimens collected every 4 or 8 hours.
  Measure of mesor (ng)
Objective sleep quality | 15 days
  Measure of sleep latency assessed by sleep log
Objective sleep quality | 15 days
  Measure of sleep latency assessed by actigraphy
Objective sleep quality | 15 days
  Measure of sleep efficiency
  = total sleep / bedtime assessed by sleep log
Objective sleep quality | 15 days
  Measure of sleep efficiency
  = total sleep / bedtime assessed by actigraphy
Objective sleep quality | 15 days
  Measure of fragmentation index assessed by sleep log
Objective sleep quality | 15 days
  Measure of fragmentation index assessed by actigraphy
Objective sleep quality | 15 days
  Measure of intra-sleep wakefulness assessed by sleep log
Objective sleep quality | 15 days
  Measure of intra-sleep wakefulness assessed by actigraphy
Objective sleep duration | 15 days
  duration of sleep assessed by actigraphy
Excessive daytime sleepiness | at day 1
  This outcome will be assessed by the Epworth sleepiness Scale
Asthenia | at day 1
  This outcome will be assessed by the Pichot asthenia scale
Insomnia severity | at day 1
  This outcome will be assessed by the Insomnia Severity Index
Anxiety | at day 1
  This outcome will be assessed by the Hospital Anxiety and Depression scale
Depression | at day 1
  This outcome will be assessed by the Hospital Anxiety and Depression scale
Vigilance at awakening | at day 2, 8 and 13
  This outcome will be assessed by the Karolinska scale
Sleep subjective quality | at day 2, 8 and 13
  This outcome will be assessed by the St Mary Hospital Questionary
Chronotype | at day 1
  This outcome will be assessed by the Horne and Ostberg Questionary
Light exposition | 15 days
  This outcome will be assessed by the actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Laure Peter Derex, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix-Rousse Hospital, Lyon, France